CLINICAL TRIAL: NCT01247532
Title: Pilot Study of Mindfulness-Based Stress Reduction for Patients With Persistent Cancer-Related Fatigue
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Walther Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Kurt Kroenke, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-01 Study 1003-02B; R25CA117865-01A11 (Other Grant/Funding Number: NCI); R25CA117865-01 (NIH)
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Cancer; Fatigue
Keywords: Cancer; Fatigue; Mindfulness; Meditation; Neoplasms
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Waitlist (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction - Cancer-Related Fatigue

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction - Cancer-Related Fatigue — 7 week 2 hour class
  Other Names: MBSR

SUMMARY:
The purposes of the proposed study are (1) to collect data on the feasibility of offering Mindfulness-Based Stress Reduction (MBSR) as an intervention to reduce fatigue and psychological distress in cancer patients who are not in active treatment for their cancer and (2) to estimate effect sizes of the intervention for fatigue, depression, anxiety, and sleep disturbance. The investigators also will obtain preliminary effect sizes of the degree to which the intervention increases mindfulness, and the investigators will evaluate dosage effects. Findings will suggest whether a future randomized controlled trial with cancer-related fatigue (CRF) as the primary outcome is feasible and warranted.

Participants will be randomly assigned to either the MBSR intervention arm or to a wait-list control arm. The MBSR intervention will consist of a weekly 2-hour class to be held for seven consecutive weeks in the Indiana University Simon Cancer Center Pavilion; the class on week six will be extended to a 3-hour "retreat." Participants will be invited to engage in daily home practice of meditation and other mindfulness exercises. All participants will complete a series of self-report questionnaires prior to the start of the classes, immediately following the end of classes, and 1 month after the class ends. Those in the intervention arm will begin the MBSR class the week after enrollment; the control group will be offered the same 7-week program after 1-month post-intervention follow-up assessments are completed-approximately 13 weeks after enrollment.

Primary Aim 1: Obtain preliminary RCT effect sizes for changes in fatigue of an MBSR treatment group compared to a wait-list control group.

Hypothesis 1: Immediately post-intervention (T2), improvements in fatigue compared to pre-intervention (T1) will be greater in the treatment group than the control group.

Hypothesis 2: At 1 month post intervention (T3), improvements in fatigue compared to pre-intervention (T1) will be greater in the treatment group than improvements in the control group.

DETAILED DESCRIPTION:
Secondary Aim 1: Obtain preliminary randomized controlled trial (RCT) effect sizes for changes in depression, anxiety, and sleep disturbance of an MBSR treatment group compared to a wait-list control group.

Hypothesis 1: Immediately post-intervention (T2), improvements in depression, anxiety, and sleep compared to pre-intervention (T1) will be greater in the treatment group than the control group.

Secondary Aim 2: Obtain preliminary effect sizes of the degree to which the intervention increases mindfulness and of the relationship of mindfulness with fatigue, depression, anxiety, and sleep disturbance.

Hypothesis 1: At T2 and 30-days post-intervention (T3), improvements in mindfulness compared to pre-intervention (T1) will be greater in the treatment group than in the control group.

Hypothesis 2: Degree of mindfulness will be negatively correlated with fatigue, depression, anxiety, and sleep disturbance at all time-points.

Secondary Aim 3: Evaluate the feasibility of recruiting fatigued cancer patients to participate in MBSR-CRF, as well as the acceptability and dosage effects of MBSR-CRF.

Hypothesis 1: At least 30% of patients who meet study criteria will choose to enroll in the proposed study.

Hypothesis 2: The MBSR intervention protocol will demonstrate feasibility in that (1) at least 70% of participants will attend at least 4 of the 7 scheduled classes, and (2) at least 70% of participants will practice mindfulness at least 60 minutes per week.

Hypothesis 3: Class attendance and hours of mindfulness practice per week will be positively associated as indicated by correlation effect sizes with improvements in both the process variable (degree of mindfulness) as well as the primary outcome variable (i.e., fatigue) and secondary outcome variables (i.e., depression, anxiety, and sleep disturbance).

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be eligible to participate based on the following criteria:

  1. they have a cancer diagnosis
  2. are age 18 or older
  3. have clinically significant cancer-related fatigue (CRF) that has persisted for the previous 8 weeks or longer. Clinically significant CRF will be defined by a cutoff mean score of ≥ 4 across the 3-item Fatigue Symptom Inventory severity composite.

Exclusion Criteria:

* Participants will be excluded based on the following criteria:

  1. chemotherapy, biologic response modifiers, radiation therapy, or surgery in prior 3 months
  2. enrollment in hospice care
  3. severe hearing impairment
  4. severe depression (PHQ-8 ≥ 15)
  5. past participation in a mindfulness meditation class
  6. incapable of reading and writing English. Each of these characteristics will be assessed as part of the eligibility screening interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Fatigue Symptom Inventory Interference Subscale | Last 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Kroenke, MD, Principal Investigator — Indiana University School of Medicine; Shelley Johns, PsyD, Study Director — Indiana University School of Medicine